CLINICAL TRIAL: NCT04441619
Title: Mechanisms and Modulation of Pain Modulatory Capacity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB20190295 3-N; R01AR073745-01A1 (NIH)
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: This is a mechanistic observational study
Who Masked: Outcomes Assessor
Masking Description: Assessments will be performed by an investigator who is not aware of the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repeated exposure (Active Comparator): Participants will complete four exercise sessions designed to induce delayed onset muscle soreness in the biceps
  Interventions: Behavioral: Delayed onset muscle soreness.
- Single exposure (Active Comparator): Participants will complete one exercise session designed to induce delayed onset muscle soreness
  Interventions: Behavioral: Delayed onset muscle soreness.
- Natural history (No Intervention): Participants will complete all sensory testing and imaging but not perform any exercise sessions.

INTERVENTIONS:
Behavioral: Delayed onset muscle soreness. — Participants will perform a fatiguing exercise protocol for the upper extremity (biceps muscles)
  Arms: Repeated exposure; Single exposure

SUMMARY:
This project proposes to understand the sources of pain variability, and demonstrate that pain variability represents fluctuation in natural pain management. The project further proposes to determine if endogenous capacity to modulate pain can be trained to maximize their body's ability to manage pain, much as the way in which athletic performance can be trained.

DETAILED DESCRIPTION:
Many physiological systems (bioenergy, immune etc.) involve feedback mechanisms to respond to challenges, with increased output or capacity for adaptive change. A similar process is plausible for pain modulation where previous successful pain experience and resolution suggests a pain modulatory system with adaptive capacity. The proposed research examines how a musculoskeletal training program modulates pain response in people with fibromyalgia compared to healthy individuals. Previous research suggests that moderate-high level exercise is associated with attenuation of pain sensitivity and clinical pain intensity in healthy individuals. The proposal seeks to extend findings from previous research and examine how repeated exposure and subsequent adaptations to musculoskeletal pain over time influence pain modulation (PMC). The first outcome is that people with fibromyalgia (FM) will have PMC trainability similar to asymptomatic controls, with the obvious implications for clinical application. The second outcome is that FM patients will demonstrate a deficit in PMC trainability. This outcome will represent an important diagnostic sign, and guide research to additional mechanistic investigation. The third outcome is that impaired or lessened PMC trainability is evident in FM patients and this variability can be explored as an individual difference with clinical implications. The theoretical fourth potential outcome is sensitization in FM patients, however pilot data show that DOMS resolves within the same relative time window as controls. Though not hypothesized, the data and design will allow for examination of this possibility. One potential conclusion from these projects could be that FM arises from an inability to enter a recovery period within which PMC could adapt and increase resilience. The proposal will be able to address at least some of the potential for this inability to recover.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic people (ie no current pain conditions)
* Participants with widespread muscle pain (WMP) aged 18 years of age and older
* Participants with WMP must meet the ACR (2010) diagnostic criteria of multiple regions of muscle pain
* The asymptomatic group will be free of current wrist/hand, elbow, or shoulder pain and chronic pain conditions (eg irritable bowel syndrome, FM)

Exclusion Criteria:

1. Participation in a conditioning program specific to the biceps in the past 6 months
2. Any report of wrist/hand, elbow, or shoulder pain in the last 3 months
3. Any chronic medical conditions that may affect pain perception (e.g., diabetes, high blood pressure), kidney dysfunction, muscle damage, or major psychiatric disorder
4. Use of any intervention (including but not limited to medication, massage, and stretching) for symptoms induced by pain training for the duration of the study
5. Positive result on pre-MRI metal screening or pregnancy test due to contraindication for the MRI environment.
6. Any participant with ferromagnetic metal in the head, neck, or abdominal cavity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline up to 10 weeks
  Pain during movement and pain at rest using the visual analog scale (VAS). Scores are recorded every day by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
Change in thermal quantitative sensory testing | Baseline up to 10 weeks
  Thermal pain thresholds and suprathreshold responses will be collected using a numeric rating scale anchored 0 "no pain" and 10 "worst pain imaginable". Change will be calculated using simple change scores and more complex multi-level modeling.
Change in pressure quantitative sensory testing | Baseline up to 10 weeks
  Pressure pain threshold will be collected using a numeric rating scale anchored 0 "no pain" and 10 "worst pain imaginable". Change will be calculated using simple change scores and more complex multi-level modeling.

SECONDARY OUTCOMES:
Cortical network connectivity | Baseline up to 10 weeks
  Functional magnetic resonance imaging of regional connectivity among pain-related brain regions

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Robinson, PhD, Principal Investigator — University of Florida
Locations (1):
- Unversity of Florida, Gainesville, Florida, United States